CLINICAL TRIAL: NCT04653779
Title: A Multi-center, Open-label, Single-arm, Phase IV Clinical Trial to Evaluate the Preference Regarding Convenience of Medication, Efficacy and Safety After Switching to SUGAMET®XR Tablet 5/1000mg in Patients With Type 2 Diabetes and Renal Diseases
Brief Title: A Clinical Trial to Evaluate the Preference Regarding Convenience of Medication and Efficacy/Safety of SUGAMET®XR Tablet 5/1000mg
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA1229_01_DM_IV
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 2; Renal Disease; Diabetes Mellitus; Metabolic Disease; Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Diseases; Diabetes Mellitus; Metabolic Diseases; Endocrine System Diseases | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): Patients receive Evogliptin 5mg/Metformin 1000mg once a day
  Interventions: Drug: Evogliptin 5mg/Metformin 1000mg

INTERVENTIONS:
Drug: Evogliptin 5mg/Metformin 1000mg — Size reduction of a tablet formulation
  Other Names: SUGAMET®XR tablet 5/1000mg

SUMMARY:
Multi-center, open-label, single arm study to Evaluate the preference regarding convenience of medication, efficacy and safety of Sugamet XR tab. 5/1000mg in patients with Type 2 diabetes and renal diseases

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥60 years
* Subjects with type 2 diabetes mellitus
* Subjects treated with DPP-4 inhibitor and 1,000mg/day dose of metformin 1T/qd for at least 8 weeks prior to screening
* Subjects with HbA1c≤7.5% at screening
* Subjects with 45mL/min/1.73m2≤eGFR≤90mL/min/1.73m2 at screening
* Subjects with fasting glucose≤200 at screening
* Subjects with 18.5kg/m2≤BMI≤40kg/m2 at screening

Exclusion Criteria:

* Patients with type 1 diabetes mellitus, secondary diabetes mellitus or gestational diabetes mellitus
* ESRD or Patients who have kidney dialysis
* Subjects with ALT and AST 3 times or higher than upper normal range

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
The preference regarding convenience of medication | 12 weeks
  Looking back on the experience of participating in the study, which would you prefer, any of the existing DPP-4 inhibitor/metformin 1000mg sustained-release combination drug or the SugarMet® sustained-release tablet 5/1000mg?

SECONDARY OUTCOMES:
Change from baseline in HbA1c (%) After 12 weeks | 12 weeks
Change from baseline in HbA1C response rate(%) After 12 weeks | 12 weeks
Change from baseline in Glycated albumin After 12 weeks | 12 weeks
Change from baseline in e-GFR After 12 weeks | 12 weeks
Change from baseline in UACR After 12 weeks | 12 weeks
  Urine Albumin-to-Creatinin Ratio
Change from baseline in HbA1c (%) After 12 weeks NAG | 12 weeks
  N-Acetyl-Glucosaminidase
Change from baseline in Nephrin After 12 weeks | 12 weeks
Change from baseline in Cystatin-C After 12 weeks | 12 weeks
TSQM-9 scores | 12 weeks
  Treatment Satisfaction Questionnaire for Medication-9 scores, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Suncheonhyang Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Se-jong hospital, Bucheon-si, Gyeonggi-do